CLINICAL TRIAL: NCT04992143
Title: The Efficacy and Safety of TACE Combined With Tilelizumab and Sorafenib in Treating BCLC Stage C HCC Patients: a Single-center, Single-arm, Prospective Clinical Study
Brief Title: TACE+Tilelizumab+Sorafenib in the Treatment of BCLC Stage C HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEPIC2004
Record Dates: First submitted 2021-08-01; First posted 2021-08-05 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: BCLC Stage C Hepatocellular Carcinoma
Keywords: BCLC Stage C; Hepatocellular Carcinoma; Transarterial Chemoembolization; Sorafenib; Tilelizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE combined Tilelizumab and Sorafenib (Experimental): TACE first combined Tilelizumab(240mg/3wks ivgtt） and Sorafenib （800mg/day orally)
  Interventions: Procedure: TACE; Drug: Tilelizumab; Drug: Sorafenib

INTERVENTIONS:
Procedure: TACE — TACE first ,and more TACE could be performed when it is necessary.
Drug: Tilelizumab — Tilelizumab 240mg per 3weeks ivgtt within 1 week after the first TACE
Drug: Sorafenib — Sorafenib should be administered 400 mg twice /day orally within 1 week after the first TACE

SUMMARY:
According to the BCLC staging system treatment recommendation, systemic treatment is recommended for patients in BCLC stage C, and TACE and systemic treatment are recommended for patients in this stage. Studies have shown that TACE combined with sorafenib therapy has shown effectiveness in the treatment of advanced liver cancer, and PD-1 inhibitors have also shown effectiveness in the treatment of advanced liver cancer. Therefore, in order to improve the survival benefit of BCLC stage C liver cancer patients, this clinical study was designed to evaluate the effectiveness and safety of TACE combined with sorafenib and tislelizumab in the treatment of BCLC stage C liver cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Child-Pugh score≤ 7
* HCC diagnosed by biopsy or by the noninvasive criteria of the Chinese Liver Cancer Guideline 2019
* the primary HCC being in BCLC C stage according to NCCN guideline
* No previous systemic therapy for HCC

Exclusion Criteria:

* Diffuse HCC
* Uncontrolled ascites of hepatic encephalopathy
* Prior liver transplantation
* Positive for human immunodeficiency virus
* Active gastric or duodenal ulcer
* Other uncontrolled comorbidities or malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
1-year survival rate | at 1 year after enrolled
  1-year survival rate assessed by Kaplan-Meier analysis

SECONDARY OUTCOMES:
Time to progression | at 12 weeks and up to 2 years after enrolled
  Time to progression assessed by independent radiologic review according to mRECIST criteria
Progression free survival | at 12 weeks and up to 2 years after enrolled
  Progression free survival assessed by independent radiologic review according to mRECIST criteria
Objective response rate | at 12 weeks and up to 2 years after enrolled
  Objective response rate assessed by independent radiologic review according to mRECIST criteria
Disease control rate | at 12 weeks and up to 2 years after enrolled
  Disease control rate assessed by independent radiologic review according to mRECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jun-hui Sun, MD,PH.D, Study Director — First Affiliated Hospital of Zhejiang University
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No